CLINICAL TRIAL: NCT06092242
Title: The Efficacy and Safety of TAS-102(Suyuan) Combined With Bevacizumab as First-line Therapy in Patients With Advanced Colorectal Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The Second Affiliated Hospital of Shandong First Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MT-006
Record Dates: First submitted 2023-10-14; First posted 2023-10-23 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Colorectal Cancer
Keywords: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Bevacizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TAS-102 combined with bevacizumab (Experimental)
  Interventions: Drug: Tas-102(Suyuan) combined with bevacizumab

INTERVENTIONS:
Drug: Tas-102(Suyuan) combined with bevacizumab — Tas-102: po 35 mg/m2, bid, d1-5, d8-12, Q4 wks; bevacizumab: intravenous drip 5 mg/kg, D1, D15, Q4 wks.

SUMMARY:
To evaluate the efficacy and safety of TAS-102 combined with bevacizumab as first-line therapy in patients with advanced colorectal cancer who could not tolerate or did not receive combined chemotherapy

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years
2. Life expectancy of at least 3 months
3. Definitive histological or cytological evidence of adenocarcinoma of the colon or rectum;
4. Patients who had not previously received first-line chemotherapy or targeted therapy for metastatic colorectal cancer, or who had received adjuvant chemotherapy after radical resection and had relapsed 12 months after completion of adjuvant chemotherapy;
5. Patients who can not or can not tolerate combination chemotherapy.
6. ECOG performance status was PS ≤2;
7. According to RECIST Version 1.1, at least 1 measurable metastatic lesion was present;
8. Appropriate organ function according to laboratory test values obtained within 7 days prior to administration of the study drug on Day 1 of Cycle 1.

   A .The hemoglobin value was more than 90 g/L. B. The absolute neutrophil count was > 1.500 MM3. C. Platelet count was > GT; 100,000/mm (> GT; 100 * 10 ° L) . D. Total serum bilirubin was 1.5 x upper limit of normal (ULN) . E.Don't L-aspartic Acid aminotransferase (asgot) and endolaminic aminotransferase (Alt SGPT)≤2.5 x upper limit of normal (ULN) , and AST and ALT ≤5 x ULN if abnormal liver function is due to basal liver metastasis.

   F. Serum creatinine ≤1.5 x upper limit of normal (ULN) or creatinine clearance ≥50 ml/min;.

   G.Adequate coagulation: international standard ratio (INR) or prothrombin time (PT)≤1.5 times the upper limit of normal;. Urine or serum pregnancy tests were negative within 7 days of randomization.
9. Women at risk of pregnancy must agree to use adequate contraception during the study until 6 months after the cessation of the study drug; Men had to agree to use adequate contraception during the study until six months after the study drug was discontinued.
10. Willing and able to follow research protocols and visit plans.

Exclusion Criteria:

1. The existence of serious diseases and serious medical conditions, this includes, but is not limited to, the following:

1. the presence of other active malignancies at the same time, excluding those that have not been diagnosed for more than 5 years or are considered curable with adequate treatment,
2. the known presence of brain or pial metastases,
3. systemic active infection (ie, infection leading to body temperature ≥38 ° C-RRB- ,
4. clinically significant intestinal obstruction, pulmonary fibrosis, renal failure, liver failure, or symptomatic cerebrovascular disease,
5. uncontrolled diabetes;
6. patients who have experienced any arterial thrombosis, embolism, or ischemic or hemorrhagic disease in the last 6 months and have not improved after appropriate treatment, such as unstable myocardial infarction, unstable angina, cerebrovascular accident after treatment,
7. severe/unstable angina, NYHA Class III or IV symptomatic congestive heart failure,
8. clinically significant gastrointestinal bleeding,
9. known presence of human immunodeficiency virus (HIV) or acquired conventional immunodeficiency syndrome (AIDS)-related disease, or active hepatitis B or C,
10. presence of psychiatric disorders that may increase the risk of participating in the study or taking research drugs, or that may interfere with the interpretation of the study results;
11. patients with grade 2 or more hypertension before treatment who had not improved or were unstable with antihypertensive drugs,
12. patients with nephrotic syndrome or with proteinuria ≥2 + or more before treatment who had not improved or were unstable after treatment, 13-RRB- patients with a history of gastrointestinal perforation in the last 6 months,
13. patients with Hypertensive crisis hypertensive encephalopathy. 2.Any of the following treatments were performed within a specific time frame prior to study drug administration,

1）major surgery (laparotomy, thoracotomy, and evisceration by laparoscopy) was performed within the previous 4 weeks. Switch surgery was not included) ; 2) had received extended-range radiotherapy within the previous 4 weeks or had received limited-range radiotherapy within the previous 2 weeks; 3) had received any investigational medication within the previous 4 weeks. 3. Neurotoxicity of CTCAE grade 2 or above that has not subsided as a result of adjuvant therapy, 4. A pregnant or lactating woman. 5. The researchers did not consider it appropriate to enter the study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-10-15 (Estimated); Primary Completion 2025-10-15 (Estimated); Study Completion 2027-10-15 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival | 2 years
  The length of time during and after the treatment of a disease, such as cancer, that a patient lives with the disease but it does not get worse

SECONDARY OUTCOMES:
Overall Survival | 3 year
  Time from randomization to death from any cause
Objective Response Rate | 2 year
  It refers to the proportion of patients (mainly solid tumors) whose tumor has shrunk to a certain extent and remained there for a certain period of time, including Complete Response (CR) and Partial Response (PR)
Quality of life score | 3 year
  Quantitative scoring system for patients' self-subjective self-assessment of current symptom tolerance

CONTACTS AND LOCATIONS:
Overall Officials: Haiyan Liu, Principal Investigator — The Second Affiliated Hospital of Shandong First Medical University
Locations (1):
- The Second Affiliated Hospital of Shandong First Medical University, Tai’an, Shandong, China